CLINICAL TRIAL: NCT00533611
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Tolerability and Effect of MK0524A on Niacin-Induced Acute Flushing in Lipid Clinic Patients
Brief Title: Effect of MK0524A on Flushing Caused by Niacin (0524A-056)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-056; MK0524A-056; 2007_604
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Flushing
MeSH Terms: conditions — Flushing | interventions — Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0524A, /Duration of Treatment : 4 Weeks
Drug: Comparator : niacin /Duration of Treatment : 1 Weeks

SUMMARY:
The primary objective of the study is to assess the effects of MK0524A in reducing flushing associated with niacin.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female between 18 and 70 years of age
* Females of reproductive potential must agree to take acceptable contraceptive precautions for the duration of the study

Exclusion Criteria:

* Patient has a history of hypersensitivity to niacin or niacin-containing products
* Patient is currently experiencing menopausal hot flashes
* Patient consumes more than 2 alcoholic beverages per day
* Patient has poorly controlled Type 1 or Type 2 diabetes mellitus
* Patient engages in vigorous exercise or an aggressive diet regimen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330
Dates: Start 2007-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
MK-0524A produces less flushing during the acute dosing period than niacin extended-release as measured by maximum Global Flushing Severity Score (GFSS) categorized as none/mild, moderate, severe, extreme. | Over 1 week

SECONDARY OUTCOMES:
MK-0524A produces less flushing during the acute dosing period than niacin extended-release as measured by (a) maximum daily GFSS; and (b) percentage of patients with a maximum GFSS =4 (moderate or greater). | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Kush D, Hu DY, Ye P, Kim HS, Chen E, Sirah W, McCrary Sisk C, Paolini JF, Maccubbin D. Flushing profile of extended-release niacin/laropiprant at initiation of therapy in Asian lipid clinic patients. Cardiology. 2009;114(3):192-8. doi: 10.1159/000228585. Epub 2009 Jul 15. PMID 19602880
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html